CLINICAL TRIAL: NCT03292198
Title: Treatment Indications for Breast Cancer-related Subclinical Lymphedema Identified Through a Bioimpedance Surveillance Model
Brief Title: Subclinical Lymphedema Treatment Study
Acronym: SLT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Collaborators: ImpediMed Limited (Industry)
Responsible Party: Principal Investigator, Megan Klote, Doctor of Physical Therapy, Certified Lymphedema Therapist - LANA, Mercy Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1070741-1
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer-related Subclinical Lymphedema
Keywords: Subclinical lymphedema; bioimpedance; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compression Group (Active Comparator): Subjects in the Compression Group will wear 20-30 mmHg sleeves and gauntlets daily for a maximum of 4 weeks. L-dex will be performed at the end of each week. If the L-dex score has reversed back into normal range, intervention (garment wearing) will be discontinued and the subject will resume the surveillance schedule of screenings. If the L-dex score is still abnormal, garment wearing continues. If L-dex score is abnormal even at the end of the 4 weeks, the subject will be removed from the study and referred to standard lymphedema therapy.
  An abnormal L-dex is defined by 7 or more units change compared to the subject's pre-surgical baseline.
  Interventions: Other: 20-30 mmHg compression sleeve and gauntlet
- Therapy Group (Experimental): Subjects in the Therapy Group will wear 20-30 mmHg sleeves and gauntlets daily and receive Manual Lymphatic Drainage 3x/week for a maximum of 4 weeks. L-dex will be performed at the end of each week. If the L-dex score has reversed back into normal range, intervention will be discontinued and the subject will resume the surveillance schedule of screenings. If the L-dex score is abnormal, intervention continues. If L-dex score is abnormal even at the end of the 4 weeks, the subject will be removed from the study and referred to standard lymphedema therapy.
  An abnormal L-dex is defined by 7 or more units change compared to the subject's pre-surgical baseline.
  Interventions: Other: 20-30 mmHg compression sleeve and gauntlet; Other: Manual Lymphatic Drainage

INTERVENTIONS:
Other: 20-30 mmHg compression sleeve and gauntlet — Compression garments are Juzo Soft, circular knit. Most will be off-the-shelf sizing, but custom when necessary.
  Garment fittings will be performed by Certified Lymphedema Therapists.
Other: Manual Lymphatic Drainage — Manual Lymphatic Drainage (MLD) is a gentle skin-stretch massage that stimulates the lymphatic system and assists in creating collateral drainage pathways out of non-intact (damaged) lymphatic territories. MLD is a critical part of Complete Decongestive Therapy (CDT), which is accepted as the international standard of care in the treatment of lymphedema.
  The MLD sessions will be performed by 2 Certified Lymphedema Therapists, Megan Klote and Sarah Stolker, both trained through the Norton School of Lymphatic Therapy. The therapists have completed reliability meetings regarding MLD sequencing and techniques.
  Other Names: MLD
  Arms: Therapy Group

SUMMARY:
Primary Objective

* To compare the effectiveness of 2 treatment protocols for patients with breast cancer-related subclinical lymphedema identified through bioimpedance spectroscopy, L-dex scores

Secondary Objectives

* To determine the necessary duration of intervention to reverse L-dex scores back to a normal range in patients with breast cancer-related subclinical lymphedema
* To determine the time elapsed post-surgically to the development of subclinical lymphedema identified by bioimpedance spectroscopy, L-dex scores
* To identify risk factors for the development of subclinical lymphedema in patients with breast cancer
* To identify factors associated with the progression to clinical lymphedema following treatment of subclinical lymphedema as identified by bioimpedance spectroscopy, L-dex scores

Women with breast cancer diagnoses and planned axillary lymph node procedures will receive pre-operative screening of arm volume with bioimpedance, which will capture baseline measurements. Then, subjects will undergo periodic screenings for the first 3 years following surgery. If a significant change in volume compared to baseline is detected with bioimpedance, subjects will be randomized to 1 of 2 treatment groups. The outcomes of 2 treatment protocols will be compared. Additionally, subjects will be screened each week during their treatment interventions to determine the necessary quantity of intervention before L-dex scores normalize.

DETAILED DESCRIPTION:
Lymphedema is an accumulation of fluid in the interstitial tissues resulting from an impairment of the normal lymphatic drainage of the affected region. Lymphedema is often a side effect of breast cancer treatments such as axillary lymph node surgery and radiation, as these procedures are damaging to the lymphatic structures. Due to poor awareness of the condition, minimal education is given to patients about their risk for lymphedema as a result of cancer treatments. With inconsistent diagnostic methods, many cases of breast cancer-related lymphedema are diagnosed after the condition has progressed to its irreversible and chronic form, i.e. clinical lymphedema.

Bioimpedance spectroscopy (BIS) uses a low frequency electrical current to assess extracellular fluid of the limbs. BIS has proven to be a sensitive and specific tool for detecting subclinical lymphedema (Stage 0) and has been validated in its use within a surveillance model. Recent literature supports the use of a surveillance model to identify breast cancer-related subclinical lymphedema to allow for early intervention and improved patient outcomes.

Despite the growing body of evidence supporting the importance of early identification of lymphedema in the subclinical stage, there is limited evidence to guide treatment of this patient population. Treatment parameters for subclinical lymphedema stem primarily from a study by Stout et al. indicating that a short compression trial (mean duration of 4.4 weeks) of 20-30 mmHg garments effectively treated subclinical lymphedema identified by perometry by preventing progression to late-stage lymphedema.

Surveillance of arm volume will be performed using bioimpedance spectroscopy (BIS) testing with the Impedimed® L-dex U400. Subjects will receive BIS testing (1) pre-operatively, (2) post-operatively at 6 weeks, (3) 3 months, (4) 6 months, (5) 12 months, (6) 18 months, (7) 24 months, and (8) 36 months. The outcome measure will be the L-dex score.

Only subjects who have an abnormal result will be enrolled in the experimental portion of the study. If an L-dex score is abnormal (defined by a change of +7 units from her pre-operative baseline), the subject is determined to exhibit subclinical lymphedema. As a result, these subjects will be randomized into one of two intervention groups. The group receiving only compression intervention will be referred to as the compression group (CG). The group receiving Manual Lymphatic Drainage (MLD) and compression will be referred to as the therapy group (TG).

Subjects will be followed through screenings for a maximum of 3 years post-surgically.

The investigators hope that this study will take the next step in the surveillance model by answering questions about how patients with subclinical lymphedema should be clinically managed.

ELIGIBILITY:
Inclusion Criteria:

New diagnosis of breast cancer, Female, 18 years of age or older, Upcoming unilateral axillary lymph node procedure (biopsy or dissection), Able to provide informed consent

Exclusion Criteria:

Pre-existing diagnosis of lymphedema, as diagnosed by physician, History of axillary lymph node procedure, including biopsy, dissection, or radiation to, Pregnancy, Pacemaker or other implanted electrical device, Stage 4-5 kidney disease, Severe liver disease, Active infection, Acute Deep Vein Thrombosis, Unmanaged congestive heart failure or a cardiac event in the past 6 months, Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
L-dex scores | 3 years post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Megan T Klote, DPT, CLT-LANA, Principal Investigator — Mercy Research
Locations (1):
- Mercy David C. Pratt Cancer Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No